CLINICAL TRIAL: NCT05585112
Title: Comparative Study of Articaine 4% Versus Lidocaine 2% in Local Anesthesia and Permanent Maxillary First Molars Affected by MIH.
Brief Title: Articaine 4% Versus Lidocaine 2% for Local Anesthesia of MIH-affected Maxillary Molars
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Tishreen U _Local anesthesia
Record Dates: First submitted 2022-10-15; First posted 2022-10-18 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2022-10

CONDITIONS: Molar Incisor Hypomineralisation
Keywords: local anesthesia; Lidocaine 2%; Articaine 4%; molars
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Intervention Model Description: A randomized, controlled, crossover, Triple-blinding clinical study, Comparison of articaine 4% and lidocaine 2%
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: as neither the child/parent, the investigator who performed the anesthesia/treatment, nor the assessors were aware of the type of anesthetic solution in order to avoid bias towards one of the solutions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Lidocaine 2%) (Active Comparator): 26 children will be injected with 1 ml of lidocaine 2% with epinephrine
  Interventions: Drug: Lidocaine 2%
- B (Articaine 4%) (Experimental): 26 children will be injected with 1 ml of Articaine 4% with epinephrine.
  Interventions: Drug: Articaine 4%

INTERVENTIONS:
Drug: Lidocaine 2% — The child will be injected with lidocaine 2%,after that the treatment will be completed , Pain during injection and treatment will be assessed using the FLACC scale and pain after injection and treatment will be evaluated using the Wong-Baker faces pain rating scale
  Other Names: A
  Arms: A (Lidocaine 2%)
Drug: Articaine 4% — The child will be injected with 4% Articaine, after that the treatment will be completed , Pain during injection and treatment will be assessed using the FLACC scale and Wong-Baker faces pain rating scale
  Other Names: B
  Arms: B (Articaine 4%)

SUMMARY:
Comparison of injection pain with lidocaine and articaine. Comparison of the efficacy of lidocaine and articaine during treatment of MIH- maxillary molars.

Design: A randomized, controlled, crossover, Triple-blinding clinical study including twenty six cooperative children, aged 6-12years old

DETAILED DESCRIPTION:
Background and Aims: Some dentists have difficulty obtaining effective anesthesia when treating MIH molars.

There are no studies comparing the effectiveness of lidocaine and articaine in MIH-maxillary molars.

Design: A randomized, controlled, crossover, Triple-blinding clinical study including twenty six cooperative children , aged 6-12 years old. Each child was randomly assigned to either articaine 4% or lidocaine 2% in their first session with the second solution being used at the second session.

ELIGIBILITY:
Inclusion Criteria:

* Absolute positive or positive behavior according to the Frankel Scale.
* child is not under the effect of any analgesics or sedatives and their weight was more than 20 kg.
* Healthy, both physically and mentally
* A child with a MIH-affected maxillary permanent first molar on the right and left sides .

Exclusion Criteria:

* children who are uncooperative
* allergic anesthetics used in the study
* children who show inflammation in the injection site.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-25 (Actual)

PRIMARY OUTCOMES:
injection pain | during the injection of local anesthesia procedure
  evaluated by outcome assessor using the Faces, Legs, Activity, Cry, Consolability Behavioral Pain Rating Scale ( FLACC scale ) ( a behavioral pain assessment scale which has five criteria face, legs, activity, cry, consolability ,which are each assigned a score of 0, 1 or 2.Total score of scale is summed in range 0 to 10, where: 0=relaxed and comfortable; 1-3=mild discomfort; 4-6=moderate pain; 7-10=severe pain)..
injection pain | Immediately after the injection of local anesthesia procedure
  self assessment pain by the children using Wong-Baker faces pain rating scale (a scale shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10,which represents "hurts like the worst pain imaginable" )
dental pain | during procedure
  evaluated by outcome assessor using the Faces, Legs, Activity, Cry, Consolability Behavioral Pain Rating Scale ( FLACC scale ) ( a behavioral pain assessment scale which has five criteria face, legs, activity, cry, consolability ,which are each assigned a score of 0, 1 or 2.Total score of scale is summed in range 0 to 10, where: 0=relaxed and comfortable; 1-3=mild discomfort; 4-6=moderate pain; 7-10=severe pain)..
dental pain | Immediately after treatment procedure
  self assessment pain by the children using Wong-Baker faces pain rating scale (a scale shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10,which represents "hurts like the worst pain imaginable" )

CONTACTS AND LOCATIONS:
Overall Officials: Nabih Raslan, Dr, Study Chair — Tishreen University; Mai Haidar, Dr, Principal Investigator — Tishreen University
Locations (1):
- Tishreen University, Latakia, Syria